CLINICAL TRIAL: NCT06592378
Title: Integration of an Opioid Dispensing, Monitoring, and Disposal Platform With a Hospital Pharmacy to Reduce Opioid Use by Discharged Emergency Department Patients
Brief Title: Opioid Management for Discharged Emergency Department Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Addinex Technologies, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R43DA060717-01 (NIH)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Bone Fractures
Keywords: opioids; fractures; pain
MeSH Terms: conditions — Fractures, Bone; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Control Adult (Active Comparator): Patients in this arm will be adults who undergo standard at-home acute pain management with opioids after treatment for isolated bone fracture (n=25)
  Interventions: Device: Standard Pill Bottle
- Control Child (Active Comparator): Patients in this arm will be children who undergo standard at-home acute pain management with opioids after treatment for isolated bone fracture (n=25)
  Interventions: Device: Standard Pill Bottle
- Device Adult (Experimental): Patients in this arm will be adults who undergo at-home acute pain management using the Addinex system after treatment for isolated bone fracture (n=25)
  Interventions: Device: Addinex
- Device Child (Experimental): Patients in this arm will be children who undergo at-home acute pain management using the Addinex system after treatment for isolated bone fracture (n=25)
  Interventions: Device: Addinex

INTERVENTIONS:
Device: Addinex — Medication dispensing system to control and monitor opioid use
  Arms: Device Adult; Device Child
Device: Standard Pill Bottle — Access and use of opioids in a standard pill bottle.
  Arms: Control Adult; Control Child

SUMMARY:
The goal of this study is to analyze the use of the Addinex system for opioid dispensing after ambulatory care to determine whether it will reduce opioid consumption, increase pill disposal, show variables that may predict opioid consumption, and determine whether this intervention is acceptable to patients.

DETAILED DESCRIPTION:
Prescription opioids remain a popular drug class with 143 million (M) opioid prescriptions written in 2020. In that same year, 8.7 million people (2.6% of the US population) misused prescription pain relievers, and overdose deaths from opioids continue to rise to 83,695 in 2022. Across six studies, 67% to 92% of patients prescribed opioids reported unused pills. In 2017, patients were prescribed 3.3 billion excess pills, yet no more than 9% of patients properly disposed of their unused opioids. Despite attempts to reduce overprescribing, increase disposal, and decrease diversion, these issues still contribute to increasing misuse, addiction, and overdose deaths.

Addinex Technologies has developed a novel system to reduce the use of opioids through controlling, monitoring, and disposing of excess opioids. The unique "closed-loop" system starts with clinicians prescribing opioids with the Addinex system. Addinex's partner pharmacy then fills the patented dispenser and delivers it to the patient. The patient uses the Addinex app to access each individual dose code and to obtain education and feedback. Finally, the patient returns the dispenser with any excess pills in a DEA-approved mailer to Addinex's partner disposal company. In a study with Columbia University Medical Center using the Addinex system with 30 post-surgical cancer patients, results showed 70% fewer pills used than prescribed, 60% fewer refills for the same surgeries, and an 84% excess pill disposal rate.

Addinex is now partnering with Brown Emergency Medicine and Rhode Island Hospital ("Brown") to perform a feasibility study using Addinex's system. We will conduct a clinical trial involving 100 patients with extremity fractures treated by the emergency department. Half the patients (25 adults and 25 minors) will utilize the Addinex system, while the other half will have their opioids dispensed in a standard pill bottle as the control group. Addinex's system promotes the return of medication using a pre-paid disposal mailer once patients have completed their course of treatment. The clinical study's main goals involve evaluating the system's effectiveness with patients obtaining same day treatment. This evaluation will encompass an analysis of medication consumption, disposal rates, pain levels, the impact of monitoring policies, and ensuring that the established commercial protocols function seamlessly. Ultimately, the project aims to demonstrate that the Addinex system can successfully operate within the broader hospital environment (same day and scheduled procedures), controlling and monitoring opioid usage, promoting patient well-being, and lowering costs.

ELIGIBILITY:
Inclusion Criteria:

* Ages six years and older
* Ability to swallow pills
* Isolated bone fracture
* Planned to receive opioids in the post-treatment period
* Not taking opioids daily prior to the procedure
* English or Spanish-speaking
* Able to give informed consent or a parent that can give informed consent
* Ownership of and comfort using apps on a smartphone with compatible operating system
* WIFI or cellular access
* Patient not admitted to hospital

Exclusion Criteria:

* Recent opioid use (last 30 days or 2 or more prescriptions in the past 3 months
* Impaired decisional capacity
* In police custody
* Ward of the state

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Median pill consumption | One month post treatment
  Patients are expected to consume at least 16% fewer pills/MMEs using the Addinex system as compared to the control group.

SECONDARY OUTCOMES:
Median disposal of opioids | 12 months post treatment
  Patients are expected to dispose of at least 50% of excess opioid pills using the Addinex system vs. 20% in the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital/Lifespan, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No